CLINICAL TRIAL: NCT06840717
Title: Association Between Cytokines Gene Single Nucleotide Polymorphisms and Type 2 Inflammatory Asthma in Children
Brief Title: Association Between Genetic Polymorphisms and Type 2 Asthma in Children
Acronym: SNP
Status: Recruiting | Type: Observational
Sponsor: Guangzhou Institute of Respiratory Disease (Other)
Responsible Party: Principal Investigator, LI-HONG SUN, Professor, Guangzhou Institute of Respiratory Disease
Other Study IDs: GuangzhouIRD-CLY
Record Dates: First submitted 2024-10-03; First posted 2025-02-21 (Actual); Last update posted 2025-02-21 (Actual); Status verified 2025-02

CONDITIONS: Asthma in Children; Genetic Disease; Inflammation
Keywords: cytokines; Single nucleotide polymorphism; type 2 inflammation; ashtma; Susceptibility
MeSH Terms: conditions — Genetic Diseases, Inborn; Inflammation; Disease Susceptibility

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples With DNA — For children enrolled in this study, 2ml EDTA anticoagulated whole blood was retained
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Case group: Diagnosis of asthma children
- Control group: Physical health of children

SUMMARY:
To further understand the role of gene single nucleotide polymorphism (SNP) in the occurrence of type 2 inflammation-related asthma in children by analyzing the gene single nucleotide polymorphism (SNP), lung function and type 2 inflammation indicators of children diagnosed with asthma in outpatient and inpatient. To provide a theoretical basis for the study of personalized treatment and prevention strategies for asthma.

DETAILED DESCRIPTION:
Type of study:

This was a prospective, randomized case-control design.To investigate the role of genetic single nucleotide polymorphisms (SNPs) in children with type 2 asthma, and the effects of SNPs on type 2 inflammatory markers and pulmonary function indicators.

Methods:

Children with asthma who were treated at our pediatric respiratory specialty clinic and who met the criteria for type 2 inflammation were included in the case group (Type 2 inflammation was considered to be present if any of the following conditions were present: Fraction of exhaled nitric oxide(FeNO)≥20ppb；Blood eosinophilcount≥350/ul；Percentage of sputum eosinophils>3%; Asthma is caused by inhaled allergens.). The control group is healthy children who underwent physical examination. To compare the differences of single nucleotide polymorphisms (SNPs) between children with type 2 asthma and healthy children, and to explore the risk factors of type 2 asthma.

The differences of indicators between different genotypes were compared, including type 2 inflammation indicators (including Fraction of exhaled nitric oxide(FeNO)、Blood eosinophil count、Percentage of sputum eosinophils and Serum total immunoglobulin E) and pulmonary function indicators(Forced expiratory volume in one second(FEV1)、Forced vital capacity(FVC)、Ratio of forced expiratory volume in one second to forced vital capacity(FEV1/FVC) and Peak expiratory flow(PEF)).

ELIGIBILITY:
Inclusion Criteria:

1. All children with asthma diagnosis accord with the GINA in 2023 edition;
2. Other diseases that could cause wheezing and cough were excluded, such as acute laryngitis, diphtheria, congenital airway abnormalities, and tracheal foreign bodies;
3. In front of the hospital 2 weeks without antibiotics, systemic hormone medication history;
4. There were no other complications, such as congenital heart disease, pneumonia, gastroesophageal reflux disease, muscle dysplasia, etc.

Exclusion Criteria:

1. Children who had taken immunosuppressants, antibiotics and other drugs for a long time before admission;
2. Children with primary immunodeficiency disease;
3. The children and their families failed to cooperate or refused the experimental observation.

Ages: 3 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Gender Based: Yes — There was no significant difference in the ratio of male to female between the case and control groups
Study Population: Children with asthma, aged 3-14 years, attending our hospital.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2024-01-30 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
type 2 inflammation indicators | Outpatient visits for the first time
  Fraction of exhaled nitric oxide(FeNO)、Blood eosinophil count、Percentage of sputum eosinophils and Serum total immunoglobulin E
pulmonary function indicators | Outpatient visits for the first time
  Forced expiratory volume in one second(FEV1)、Forced vital capacity(FVC)、Ratio of forced expiratory volume in one second to forced vital capacity(FEV1/FVC) and Peak expiratory flow(PEF)
single nucleotide polymorphism | Outpatient visits for the first time
  Differences in SNPs of genes detected in children's blood samples

CONTACTS AND LOCATIONS:
Locations (1):
- Guangzhou institute of respiratory disease, Guangzhou, Guangdong, China